CLINICAL TRIAL: NCT06011733
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Bimekizumab in Chinese Adult Study Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Chinese Adult Study Participants With Moderate to Severe Plaque Psoriasis
Acronym: BE SHINING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0041
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Chronic Plaque Psoriasis
Keywords: Psoriasis; PSO; Bimekizumab; Chinese Adults Study Participants
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bimekizumab (Experimental): Study participants randomized to this arm will receive bimekizumab (BKZ) dosage regimen 1 in the Initial Treatment Period (16 weeks) and switch to dosage regimen 2 and placebo to maintain the blinding in the Maintenance Treatment Period (16 weeks).
  Interventions: Other: Placebo; Drug: Bimekizumab
- placebo (Placebo Comparator): Study participants randomized to this arm will receive placebo comparator in the Initial Treatment Period (16 weeks) and switch to bimekizumab dosage regimen 1 in the Maintenance Treatment Period (16 weeks).
  Interventions: Other: Placebo; Drug: Bimekizumab

INTERVENTIONS:
Other: Placebo — Study participants will receive placebo subcutaneously at pre-specified time points in the placebo arm as comparator and in the bimekizumab arm to maintain the blinding.
Drug: Bimekizumab — Study participants will receive bimekizumab (dosage regimen 1 and 2) subcutaneously administered at pre-specified time points during the Initial and Maintenance Treatment Periods.
  Other Names: BKZ

SUMMARY:
The primary purpose of this study is to compare the efficacy of bimekizumab administered subcutaneously (sc) for 16 weeks versus placebo in the treatment of study participants with moderate to severe plaque psoriasis (PSO).

ELIGIBILITY:
Inclusion Criteria:

* Study participant is Chinese male or female ≥18 years of age
* Study participant has plaque psoriasis (PSO) for ≥6 months prior to the Screening Visit
* Study participant has Psoriasis Area and Severity Index (PASI) ≥12 and body surface area (BSA) affected by PSO ≥10% and Investigator's Global Assessment (IGA) score ≥3 on a 5-point scale.
* Study participant is a candidate for systemic PSO therapy and/or phototherapy
* Female study participants must be postmenopausal or permanently sterilized or if childbearing potential must be willing to use protocol defined highly effective method of contraception throughout the duration of the study until 17 weeks after last administration of investigational medicinal product (IMP) and have a negative pregnancy test at Screening and prior to first dose

Exclusion Criteria:

* Female study participant who is breastfeeding, pregnant, or plans to become pregnant during the study or within 17 weeks following the final dose of IMP
* Study participant has a form of PSO other than chronic plaque-type (eg, pustular, erythrodermic, guttate, or drug-induced PSO)
* Study participant has an active infection or history of infection(s) as defined in the protocol
* Study participant has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection.Study participant has a past history of active TB involving any organ system unless adequately treated and is proven to be fully recovered upon consult with a TB specialist
* Study participant has a diagnosis of inflammatory conditions other than PSO vulgaris or psoriatic arthritis (PsA)
* Study participant has presence of significant uncontrolled neuropsychiatric disorder. Study participants with history of suicide attempt within the 5 years prior to the Screening Visit must be excluded. Study participants with history of suicide attempt more than 5 years prior to the Screening Visit must be evaluated by a mental health care practitioner before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index 90 (PASI90) response at Week 16 | Week 16
  The PASI90 response assessments are based on at least 90% improvement in PASI score from Baseline. Body divided into 4 areas: head, upper extremities, trunk and lower extremities. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Investigator´s Global Assessment (IGA) 0/1 response at Week 16 | Week 16
  The IGA measures the overall psoriasis severity using a 5-point scale (0-4), where 0=clear - no signs of psoriasis; post-inflammatory hyperpigmentation may be present, 1=almost clear - no thickening; normal to pink coloration; no to minimal focal scaling, 2=mild - just detectable to mild thickening; pink to light red coloration and predominately fine scaling, 3=moderate - clearly distinguishable to moderate thickening; dull to bright red, moderate scaling and 4=severe - severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response at week 16 is defined as a score of 0 or 1 with at least a two-category improvement from Baseline.

SECONDARY OUTCOMES:
PASI75 response at Week 4 | Week 4
  The PASI75 response at Week 4 is a key secondary endpoint. PASI75 response assessments are based on at least 75% improvement in PASI score from Baseline. Body divided into 4 areas: head, upper extremities, trunk and lower extremities. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
PASI100 response at Week 16 | Week 16
  The PASI100 response at Week 16 is a key secondary endpoint. PASI100 response assessments are based on a 100% improvement in PASI score from Baseline. Body divided into 4 areas: head, upper extremities, trunk and lower extremities. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease
Patient Symptom Diary (PSD) Psoriasis Symptom and Impact Measure (P-SIM) response for itch at Week 16 | Week 16
  The PSD (P-SIM) is designed to collect data about the experience of patients with moderate to severe psoriasis related to the severity of signs, symptoms or impacts, at their worst during the past 24 hours, on a 0-10 point numeric rating scale (NRS) where 0 (no symptom/ impact) and 10 (very severe symptom/ worst impact). It consists of 14 items of which three were used as secondary endpoints: Skin pain, Itch and Scaling. Itch response is defined as a reduction from Baseline to week 16 of at least 4 points on the PSD itch score.
PSD (P-SIM) response for pain at Week 16 | Week 16
  The PSD (P-SIM) is designed to collect data about the experience of patients with moderate to severe psoriasis related to the severity of signs, symptoms or impacts, at their worst during the past 24 hours, on a 0-10 point numeric rating scale (NRS) where 0 (no symptom/ impact) and 10 (very severe symptom/ worst impact). It consists of 14 items of which three were used as secondary endpoints: Skin pain, Itch and Scaling. Pain response is defined as a reduction from Baseline to week 16 of at least 4 points on the PSD pain score.
PSD (P-SIM) response for scaling at Week 16 | Week 16
  The PSD (P-SIM) is designed to collect data about the experience of patients with moderate to severe psoriasis related to the severity of signs, symptoms or impacts, at their worst during the past 24 hours, on a 0-10 point numeric rating scale (NRS) where 0 (no symptom/ impact) and 10 (very severe symptom/ worst impact). It consists of 14 items of which three were used as secondary endpoints: Skin pain, Itch and Scaling. Scaling response is defined as a reduction from Baseline to week 16 of at least 4 points on the PSD scaling score.
Incidence of Treatment-emergent Adverse Events (TEAE)s through Week 16 | From Baseline to End of initial Treatment Period (up to Week 16)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP.
Incidence of serious TEAEs through Week 16 | From Baseline to End of initial Treatment Period (up to Week 16)
  An SAE is any untoward medical occurrence that at any dose:
  Results in death Is life-threatening Requires in patient hospitalisation or prolongation of existing hospitalisation Is a congenital anomaly or birth defect Is an infection that requires treatment with parenteral antibiotics Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of TEAEs leading to permanent discontinuation of Investigational Medicinal Product (IMP) through Week 16 | From Baseline to End of initial Treatment Period (up to Week 16)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs leading to withdrawal of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (18):
- China (18):
  - Ps0041 20023, Beijing
  - Ps0041 20247, Beijing
  - Ps0041 20306, Beijing
  - Ps0041 20117, Guangzhou
  - Ps0041 20311, Guangzhou
  - Ps0041 20313, Guangzhou
  - Ps0041 20022, Hangzhou
  - Ps0041 20193, Hangzhou
  - Ps0041 20296, Hangzhou
  - Ps0041 20312, Jinan
  - Ps0041 20318, Jinan
  - Ps0041 20310, Ningbo
  - Ps0041 20308, Shanghai
  - Ps0041 20184, Shenzhen
  - Ps0041 20136, Tianjin
  - Ps0041 20120, Wuhan
  - Ps0041 20314, Wuxi
  - Ps0041 20309, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org